CLINICAL TRIAL: NCT05908474
Title: Preliminary Pilot Exploratory Investigations Into the Effects of io Fibrewater Supplementation on Body Composition Parameters, Blood Chemistry and Cognitive, Psychological, and Behavioural Factors in Overweight Adults
Brief Title: The Effects of io Fibrewater Supplementation on Gut Health, Immunity and Metabolism in Overweight Adults
Acronym: IOFW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roehampton (Other)
Responsible Party: Principal Investigator, DR ADELE COSTABILE, Associate Professor in Health Sciences and Nutrition, University of Roehampton
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LSC 23/ 383
Record Dates: First submitted 2023-05-31; First posted 2023-06-18 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: A 30-day placebo-controlled randomised trial study in overweight adults who have not been diagnosed with Diabetes
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iowater fibre Group (Active Comparator): This exclusive blend of scientifically substantiated ingredients has been demonstrated to contribute to the reduction of body weight and aid the sustainability of weight loss by providing a healthy, hunger-free weight management system. iofibrewater, makes fibre and gut health simple and refreshing. Each 500 ml bottle of ió fibrewater provides 20%* of your recommended daily fibre intake and 100%* of your daily prebiotic fibre intake with minimal calories and carbohydrates, making us suitable for people on a variety of diets. ió fibrewater is a functional water infused with prebiotic fibre (aka prebiotics), which leads to sub-optimal gut health and often the onset of digestive disorders. By adding more prebiotic fibre to our diet, we can quickly change the environment in our gut for the better healthy living.
  Interventions: Dietary Supplement: Enriched fibre water
- Volvic Placebo control Group (Placebo Comparator): This is the equivalent placebo control water that it is matching the energy values
  Interventions: Dietary Supplement: Enriched fibre water

INTERVENTIONS:
Dietary Supplement: Enriched fibre water — Blend of scientifically substantiated ingredients has been demonstrated to contribute to the reduction of body weight and aid the sustainability of weight loss by providing a healthy, hunger-free weight management system. iofibrewater, makes fibre and gut health simple and refreshing. Each 500 ml bottle of ió fibrewater provides 20%* of your recommended daily fibre intake and 100%* of your daily prebiotic fibre intake with minimal calories and carbohydrates, making us suitable for people on a variety of diets. ió fibrewater is a functional water infused with prebiotic fibre (aka prebiotics), which leads to sub-optimal gut health and often the onset of digestive disorders. By adding more prebiotic fibre to our diet, we can quickly change the environment in our gut for the better healthy living.
  Other Names: Io fibre water

SUMMARY:
Despite availability of many alternative and conventional weight loss options, the prevalence of obesity increased from 15% in 1993 to 27 in 2015. In 2015, 68% of men and 58% of women in the UK were overweight or obese. Overweight and obesity increase the risk for comorbidities such as hypertension, dyslipidaemia, cardiovascular disease, type 2 diabetes and certain cancers. Hormonal regulation of appetite has been shown to influence body weight and body fat . Gut hormones secreted from the intestine are particularly important both in the regulation of appetite and blood glucose level, and recently the gut hormone Glucagon Like Peptide -1 (GLP-1) has been successfully targeted to treat both type 2 diabetes and obesity. Targeting the gut microbiota has been shown to influence gut hormones, in a way is likely to help treat or prevent obesity and type 2 diabetes. In past decades, considerable attention has been given to investigating the new applications of natural prebiotic polymers on gut microbiota composition. Moreover, recent trend in research indicates a bidirectional communication between the gut microbiota and the central nervous system through the microbiome-gut-brain axis (MGBA).

Therefore an in vivo intervention feeding study is proposed performed with a variety of psychological and nutritional tests aiming to compare io fibrewater with an equivalent placebo control water and also highlight both cognitive function, emotional bias and response to appetite and also metabolic profiles of the gut microbiota.

DETAILED DESCRIPTION:
Study design: A 30-day placebo-controlled randomised trial study in overweight adults who have not been diagnosed with Diabetes.

Participants: 20 participants will be invited to take part in this study. They will be randomly assigned to treatment (n=10) or control (n=10) groups, where they will consume io Fibrewater or Volvic sugar free Lemon & Lime water for 4 weeks. Both water samples (1 bottle/day) need to be taken with the meals (lunch).

ELIGIBILITY:
* Inclusion criteria

  1. Females and males, aged 18 years to 65 years
  2. BMI ≥25 kg/m2 with any of the following:

     1. IGT (blood glucose level of 7.8-11.0 mmol/L after a 2-hour oral glucose tolerance test (OGTT)), or
     2. IFG (fasting blood glucose level of 5.6-6.9 mmol/L) or
     3. impaired HbA1c (HbA1c level of 5.7%-6.4%)
  3. Not dieting within the last month
  4. not having lost >5% body weight in the previous year
  5. Not increased physical activity levels in the past 2-4 weeks or intending to modify them during the study.
  6. Understands and is willing, able and likely to comply with all study procedures and restriction including being willing to follow the nutritional advice.
  7. Able to eat most everyday foods with no current IBS symptoms.
  8. Habitually consumes three standard meals a day (i.e., breakfast, lunch, and dinner)
* Exclusion criteria Current use of prescribed medication for neuropsychiatric disorders or history of neuropsychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
Anthropometric measurements | Change in body fat percentage from baseline and after 30 days of intervention
  Body fat percentage

SECONDARY OUTCOMES:
Blood pressure | Change in blood pressure from baseline and after 30 days of intervention
  Blood pressure readings
Gastrointestinal symptoms | Change from the baseline in bowel habits including stool frequency and consistency (Bristol stool scale), stomach or intestinal bloating, abdominal pain, incidence and frequency of flatulence
  Details of bowel habits including stool frequency and consistency (Bristol stool scale), stomach or intestinal bloating, abdominal pain, incidence and frequency of flatulence
Gut microbiota composition | Change in gut microbiota composition from baseline and after 30 days of intervention
  Details on the gut microbiota composition
Fasting blood glucose via OGGT | Change in plasma blood glucose from baseline and after 30 days of intervention
  A baseline sample will be take and the participants will be asked to drink 250mL of active or the equivalent placebo water.
  • The participants will then receive a 50 g glucose drink (orally) in 250ml of water which is commonly used to evaluate pancreatic function and the rate of changes in plasma insulin and glucose (Stumvoll, 2000) and they will donate a total of 7 venous blood samples (up to 5 ml of blood samples at each time point; 30 ml maximum total) at 15, 30, 45, 60, 75, 90, and 120 minutes.
Neurocognitive and Mood Assessment | Changes in Neurocognitive and Mood Assessment from baseline and after 30 days of intervention
  Neurocognitive and Mood Assessments will take around 60 minutes, but the visits can take up to 120 mins to complete and then will be presented on Qualtrics and Inquisit.
  Qualtrics is an Experience Management (XM) platform hosted by the university of Roehampton. The exportation of results is only allowed for users who are granted an appropriate account permission, controlled by brand administrators from the university of Roehampton. Qualtrics follows General Data Protection Regulation (GDPR) and comply with applicable data privacy laws.
  Inquisit is a powerful, easy-to-use psychological measurement and experimentation tool. Inquisit is ideal for lab-based research, cognitive neuroscience, and field testing with laptops. It allows for testing of various cognitive processes including, but not limited to, attention, inhibition, working memory and decision-making.

CONTACTS AND LOCATIONS:
Overall Officials: Adele Costabile, Study Director — The University of Roehampton
Locations (1):
- Health Sciences Research Centre, Life Sciences Department, University of Roehampton, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No